CLINICAL TRIAL: NCT06756581
Title: Tolerability of Baked Dairy Protein in Eosinophilic Esophagitis Patients With Cow Milk Protein Trigger
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Oren Ledder, MD, Dr. Oren Ledder, Principal Investigator, Shaare Zedek Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EoE tolerability of baked milk
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Eosinophilic Esophagitis (EoE)
Keywords: Eosinophilic Esophagitis (EoE)
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tolerability of baked milk products in eosinophilic esophagitis patients with cow milk trigger (Experimental): Elimination of none baked cow milk from diet . Baked milk products containing diet.
  Interventions: Other: baked milk product diet

INTERVENTIONS:
Other: baked milk product diet — Elimination of none baked cow milk from diet . Baked cow milk containing diet.

SUMMARY:
Eosinophilic esophagitis (EoE) is a chronic immune mediated disease characterized by eosinophilic infiltration in esophageal epithelium and resulting in esophageal dysfunction.

While the exact pathogenesis is yet to be elucidated, EoE is considered an atopic disease. This classification is in part due to the inflammatory infiltrate of eosinophils, basophils and T-cells producing Th2 cytokines, yet it may also be triggered by environmental allergens. In addition, the rates of atopy are approximately 3 times higher in patients with EoE than in the general population. Furthermore, and most convincing, EoE is successfully managed with dietary exclusion of triggering groups in both pediatric and adult patients, further confirming the atopic nature of the disease.

The most frequent dietary trigger for EoE is milk, but there is limited data on the effect of baked dairy . Guidelines addressing the diagnosis and treatment of EoE in both children and adults have not addressed the use of baked dairy in patients with cow's milk triggered EoE.

Restrictive diets are often challenging for patients and contribute to a reduced quality of life. Some patients tolerate baked dairy products, which are less allergenic due to denaturation of proteins through heat. The potential for baked dairy to be included in the diet of milk-triggered EoE patients remains unexplored in current guidelines.

The aim of this study is to assess tolerability and safety of baked dairy in patients with EoE in whom cow's milk has been confirmed to be a trigger food for their disease.

DETAILED DESCRIPTION:
This prospective, multi-center trial will include patients with EoE diagnosed according to the accepted definitions: symptoms of esophageal dysfunction and >15 Eos/HPF on an esophageal biopsy, who were confirmed to have cow's milk as a trigger by demonstrating improvement during elimination and histologic relapse following reintroduction.

Following full informed consent of the patient / guardians, patients will be offered to join the trial to assess their tolerance to baked dairy.

Due to the theoretical risk of developing IgE-mediated allergy on prolonged food protein type restriction, RAST-testing or skin-prick testing to cow milk will be undertaken to exclude IgE-mediated sensitization prior to introduction of baked daury. In patients with positive results, candidates can elect to withdraw from the study or alternatively an allergist will be consulted to consider the appropriateness of a medically observed baked dairy challenge.

Strict compliance with milk-free diet will be re-enforced for not less than 6 weeks prior to the patient's closest routine follow-up endoscopy. Baseline symptom profile will be recorded. Baseline endoscopy with routine biopsies (defined below) will be performed as part of the routine scheduled follow-up endoscopy as recommended by guidelines, in order to confirm histologic remission of EoE. Patients with baseline esophageal inflammation will be excluded from the study. Patients in histologic remission will be commenced on bake dairy containing diet with not less than 1 daily serving.

Repeat symptom profile assessed at 6 weeks and at 12 weeks, with repeat endoscopy with routine biopsies at 12±2 weeks. If symptoms recur prior to 12 weeks, endoscopy may be moved up earlier, from 6 weeks onwards.

Patients in clinical and histologic remission at 12 weeks will be followed until week 52 with repeat scheduled endoscopy. Baked dairy consumption will be permitted during the follow-up, but not be required daily as in the first time period. A baked dairy consumption diary will be collected over the 4 weeks prior to this endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with EoE age ≤ 17.5 years at inclusion who were confirmed to have cow's milk as a trigger by demonstrating improvement during elimination and histologic relapse following reintroduction
* Verified histologic remission on milk-free diet on endoscopy prior to intervention
* Proton-pump inhibitors may be used if treatment is maintained at the same dose from the screening endoscopy throughout the trial period, and was used at the time that milk was demonstrated to be the triggering food
* Ability to consent to enrollment in the trial - legal guardians with joint consent for patients >10 years.

Exclusion Criteria:

* Patients with clinical IgE-mediated milk allergy
* Provisional exclusion: patients without a known IgE-mediated allergic reaction to milk who have a positive RAST (as per local reference range) or positive skin-prick test for cow milk or goat milk must be assessed by a certified allergist/immunologist and cleared for the trial by a supervised milk challenge.
* Use of inhaled corticosteroids for more than 5 days per month during the trial period.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Histologic remission rate following 12 weeks exposure to ingested baked dairy products | 12 weeks exposure to ingested baked dairy products
  will be assessed on biopsies collected at week 12 during upper endoscopy

SECONDARY OUTCOMES:
Symptom scores following 12 weeks exposure to ingested baked dairy | 12 weeks exposure to ingested baked dairy
  Symptom profile assessed by PEESSv2.0 at 6 weeks and at 12 weeks, with repeat endoscopy with routine biopsies at 12 weeks
Endoscopic remission rate following 12 weeks exposure to ingested baked dairy | 2 weeks exposure to ingested baked dairy
  endoscopy with routine biopsies at 12 weeks
Endoscopic improvement following 12 weeks exposure to ingested baked dairy | 12 weeks exposure to ingested baked dairy
  endoscopy with routine biopsies at 12 weeks
Safety of cow's milk challenge | 36 months
  In patients with any prior suspicion of IgE-mediated cow's milk allergy including any suspicious rash or other symptoms on previous exposure, will be referred to a pediatric immunologist for assessment and consideration of RAST test or skin-prick test, with a supervised challenge, if deemed necessary, prior to enrollment in the trial. Number of participants without a positive RAST test or skin-prick test

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided